CLINICAL TRIAL: NCT00958230
Title: An Open Arm Pilot Study to Evaluate the Safety and Performance of the dCell Vascular Patch in Reconstructive Peripheral Vascular Surgery
Brief Title: dCell Vascular Patch in Peripheral Vascular Surgery Study for CE Mark Submission
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tissue Regenix Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRL P001-09
Record Dates: First submitted 2009-08-11; First posted 2009-08-13 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2010-09

CONDITIONS: Peripheral Arterial Vascular Occlusion
Keywords: endarterectomy; dCell; Tissue Regenix Ltd; TRL; Vascular Patch; Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- dCell Vascular Patch (Experimental): This Xenograft device is manufactured from Porcine Pericardium Tissue which has been decellularised leaving a scaffold style structure for ingrowth of human endothelial cells after placement into the operative site.
  Interventions: Device: dCell Vascular Patch

INTERVENTIONS:
Device: dCell Vascular Patch — Implantation of a dCell Vascular Patch as part of an Endarterectomy

SUMMARY:
The study is designed to produce early safety and performance data in a small group of patients requiring repair of a peripheral vascular endarterectomy (incision into an artery feeding the limbs which requires a patch to repair the incision after removal of an atherosclerotic plaque that was stopping usual blood flow to the limbs).

Data is being collected to show the procedure is safe and allows for normal blood flow to be resumed.

Data will be used to facilitate CE Mark submission.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for a remote or open peripheral vascular endarterectomy
2. Lack of suitable autologous material to function as closure patch for the arteriotomy
3. Uncomplicated standard elective endarterectomy procedure (per-operative inclusion criteria)
4. Use of dCell™ Vascular Patch as arteriotomy closure material (per-operative inclusion criteria)
5. Patients between 18 and 80 years old, inclusive
6. Haemoglobin > 9 g/dL and platelet count > 100,000/mm3 prior to Day 1
7. Other haematological and biochemical parameters within a range acceptable for the administration of general anesthesia prior to Day 1
8. Ability to communicate meaningfully with investigative staff, competence to give written informed consent, and ability to comply with entire study procedures
9. Duly executed, written, informed consent obtained from patient

Exclusion Criteria:

1. Known serious allergy to contrast agent used for angiography
2. Treatment with any investigational drug or device within 60 days prior to study entry (Day 1)
3. If female and of child-bearing potential: evidence of a positive pregnancy test or a stated intention to become pregnant in the next 6-12 months
4. Patients receiving a revision of an existing graft
5. Patients demonstrating an active local or systemic infection (WBC > 15,000/mm3)
6. Any condition which in the judgment of the Investigator would preclude adequate evaluation of dCell™ Vascular Patch's safety and performance
7. Patients on vitamin K antagonists

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2009-08; Primary Completion 2010-04 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Maintenance of Arterial Patency | 6 months for CE Mark, 24 months Post Market Surveillance

SECONDARY OUTCOMES:
Complication Rate | 6 months for CE Mark, 24 months for PMS

CONTACTS AND LOCATIONS:
Overall Officials: Keith Summerhayes, BSc (Hons), Study Director — Tissue Regenix Ltd
Locations (4):
- Hungary (3):
  - Szent Imre Hospital, Budapest
  - Miskolc Hospital, Miskolc
  - Semmelweis University Hospital, Semmelweis
- Saint Elisabeth Hospital, Otrobanda, Curacao, Netherlands